CLINICAL TRIAL: NCT07251231
Title: Effectiveness of Virtual Reality in Parkinson's Disease: Impact on Balance, Fall Risk, and Cardiorespiratory Exercise Capacity.
Brief Title: Effectiveness of Virtual Reality in Parkinson's Disease: Effects on Balance, Fall Risk, and Exercise Capacity.
Acronym: Parkinson
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Borja Pérez-Domínguez, Associate Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-FIS-3990912
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Virtual Reality; Postural Balance; Frailty; Exercise Tolerance
MeSH Terms: conditions — Parkinson Disease; Frailty

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): Participants receiving an intervention through Virtual Reality
  Interventions: Other: Virtual Reality
- Conventional Rehabilitation (Active Comparator): Participants receiving conventional rehabilitation
  Interventions: Other: Conventional Rehabilitation

INTERVENTIONS:
Other: Virtual Reality — Rehabilitation through a Virtual Reality program
  Arms: Virtual Reality
Other: Conventional Rehabilitation — Rehabilitation received through conventional programs
  Arms: Conventional Rehabilitation

SUMMARY:
The goal of this clinical trial is to evaluate whether immersive virtual reality (VR)-based physiotherapy is effective in improving balance, reducing fall risk, and enhancing cardiorespiratory exercise capacity in individuals with Parkinson's disease. The main questions it aims to answer are:

Does immersive VR therapy improve postural balance more effectively than conventional physiotherapy?

Does immersive VR reduce fall risk and increase cardiorespiratory fitness compared with standard physiotherapy?

Researchers will compare an immersive VR intervention with conventional physiotherapy to determine whether VR can produce superior functional and physiological outcomes in patients with Parkinson's disease.

Participants will:

Be randomly assigned (1:1) to an experimental group (immersive VR therapy) or a control group (conventional physiotherapy).

Take part in structured physiotherapy sessions focused on balance, mobility, and functional capacity.

Undergo pre- and post-intervention assessments of balance, fall risk, cardiorespiratory exercise capacity, and quality of life.

This randomized controlled trial (RCT) with parallel assignment will include 50 participants (25 per group). Randomization will be performed using the OxMaR (Oxford Minimization and Randomization) software, which enables adaptive randomization to ensure balanced baseline characteristics between groups.

Secondary objectives include evaluating the impact of immersive VR on health-related quality of life and comparing treatment adherence between VR-based and conventional physiotherapy interventions.

DETAILED DESCRIPTION:
Neurological disorders are among the leading causes of disability worldwide, significantly affecting functional independence, mobility, and quality of life. Parkinson's disease (PD) is a progressive neurodegenerative disorder characterized by dopaminergic neuron loss in the substantia nigra, resulting in motor and non-motor symptoms that compromise multiple physiological systems. The main motor symptoms-bradykinesia, rigidity, resting tremor, and postural instability-directly impair balance and substantially increase the risk of falls. Additionally, individuals with PD often exhibit reduced cardiorespiratory fitness, which contributes to functional decline, decreased participation in daily activities, and increased caregiver burden.

Physiotherapy plays a crucial role in the comprehensive management of PD, targeting improvements in balance, mobility, motor function, and cardiorespiratory capacity to delay disability and promote autonomy. In recent years, emerging technologies have transformed conventional rehabilitation paradigms, with virtual reality (VR) gaining recognition as a promising tool for enhancing therapeutic outcomes.

Immersive VR systems provide controlled, interactive, and multisensory environments that facilitate repetitive, task-oriented motor practice with immediate sensory feedback. These features can increase motivation, engagement, and adherence to therapy, while simultaneously stimulating both motor and cognitive domains. Moreover, VR interventions may induce neuromodulation processes by activating and reorganizing neural circuits, thereby promoting neuroplasticity - a fundamental mechanism for functional recovery in neurodegenerative diseases such as PD.

Preliminary research suggests that VR-based rehabilitation can lead to measurable improvements in balance, reduction in fall risk, and enhancement of physical endurance. However, the current body of evidence remains limited by small sample sizes, heterogeneous methodologies, and a lack of direct comparisons with conventional physiotherapy. Gaps persist regarding which subgroups of PD patients benefit most, the medium- and long-term effects of VR interventions, and the neurophysiological mechanisms underlying these improvements.

This randomized controlled trial (RCT) aims to address these limitations by conducting a rigorous evaluation of an immersive VR intervention compared to standard physiotherapy in individuals with PD. A total of 50 participants will be randomly assigned (1:1) to either a VR group or a conventional physiotherapy group using the OxMaR (Oxford Minimization and Randomization) software, which employs adaptive minimization to balance baseline characteristics between groups.

The primary objective is to determine whether immersive VR therapy leads to greater improvements in postural balance, fall risk reduction, and cardiorespiratory exercise capacity compared to conventional physiotherapy. Secondary objectives include assessing changes in health-related quality of life and evaluating adherence to treatment protocols across intervention groups.

By integrating neurorehabilitation principles with immersive technology, this study aims to contribute robust scientific evidence supporting the use of VR as an effective physiotherapeutic tool for enhancing functional outcomes and overall well-being in individuals with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Age between 55 and 75 years.
* Clinical diagnosis of Parkinson's disease confirmed by a neurologist.
* Mild to moderate disease stage (Hoehn and Yahr I-III).
* Ability to understand and follow simple instructions and actively participate in the intervention.
* Signed informed consent provided before participation.

Exclusion Criteria:

* Severe cognitive impairment, defined as a Montreal Cognitive Assessment (MoCA) score < 21.
* Severe musculoskeletal comorbidities that limit mobility or prevent participation in physiotherapy sessions.
* Visual or vestibular disorders that would compromise safe use of virtual reality equipment.
* Serious medical complications during the study (e.g., acute cardiovascular events such as myocardial infarction or stroke) that may endanger the participant or interfere with treatment.
* Adverse effects related to the intervention, including severe dizziness, persistent nausea, disorientation, or headaches that prevent continuation of therapy.
* Lack of adherence to the protocol, defined as missing four or more intervention sessions without justification.
* Significant worsening of neurological status or new complications that contraindicate participation in physiotherapy.
* Surgical or medical procedures unrelated to Parkinson's disease that affect general mobility or the ability to participate in the intervention.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Balance | From baseline to 12 weeks
  Balance will be assessed using the Berg Balance Scale (BBS), a standardized and validated clinical tool widely used to evaluate static and dynamic balance in individuals with Parkinson's disease. The BBS consists of 14 functional tasks (such as standing up, reaching forward, turning, and standing on one foot), each scored on a 5-point scale ranging from 0 (unable to perform) to 4 (normal performance).
  The total score ranges from 0 to 56 points, with higher scores indicating better balance and lower fall risk. Assessments will be conducted by trained physiotherapists blinded to group allocation to ensure objectivity and minimize bias.

SECONDARY OUTCOMES:
Fall Risk and Functional Mobility | From baseline to 12 weeks
  Fall risk and functional mobility will be evaluated using two standardized clinical tests: the Timed Up and Go Test (TUG) and the Dynamic Gait Index (DGI).
  The TUG test measures the time (in seconds) it takes for a participant to stand up from a chair, walk three meters, turn, return, and sit down. Shorter times indicate better mobility and lower fall risk.
  The DGI assesses dynamic balance during walking tasks such as changing speed, turning the head, and stepping over obstacles. It includes 8 items scored from 0 to 3, with a maximum score of 24 points. Higher scores represent better gait stability and lower risk of falls.
Cardiorespiratory Exercise Capacity | From baseline to 12 weeks
  Cardiorespiratory exercise capacity will be assessed using the 6-Minute Walk Test (6MWT), a validated and widely used measure of submaximal aerobic capacity in individuals with Parkinson's disease. During the test, participants are instructed to walk as far as possible along a 30-meter corridor for six minutes at a self-paced but consistent effort level.
  The total distance walked (in meters) will be recorded as the outcome variable. Greater distances indicate improved exercise tolerance and cardiorespiratory fitness.
  All tests will be conducted under standardized conditions, with continuous supervision by trained physiotherapists to ensure safety. Participants may rest as needed, but the timer will continue running.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physiotherapy. University of Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No